CLINICAL TRIAL: NCT04632940
Title: A Phase 3, Randomized, Double-Blind, Trial of Pamrevlumab (FG-3019) or Placebo in Combination With Systemic Corticosteroids in Ambulatory Subjects With Duchenne Muscular Dystrophy (DMD)
Brief Title: Phase 3 Trial of Pamrevlumab or Placebo in Combination With Systemic Corticosteroids in Participants With Ambulatory DMD
Acronym: LELANTOS-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study did not meet its primary endpoint.
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-3019-094; 2020-000699-39 (EudraCT Number)
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy, DMD; Muscular Dystrophies; Muscular Dystrophy, Duchenne; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked | interventions — pamrevlumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pamrevlumab (Experimental): Pamrevlumab 35 milligrams (mg)/kilogram (kg) intravenously (IV) every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks
  Interventions: Drug: Pamrevlumab; Drug: Corticosteroids
- Placebo (Placebo Comparator): Matching placebo IV every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks
  Interventions: Drug: Placebo; Drug: Corticosteroids

INTERVENTIONS:
Drug: Pamrevlumab — Pamrevlumab will be administered per dose and schedule specified in the arm description.
  Other Names: FG-3019
  Arms: Pamrevlumab
Drug: Placebo — Placebo will be administered per schedule specified in the arm description.
  Arms: Placebo
Drug: Corticosteroids — Systemic deflazacort or equivalent potency of corticosteroids administered orally

SUMMARY:
To evaluate the efficacy and safety of pamrevlumab versus placebo in combination with systemic corticosteroids administered every 2 weeks in ambulatory participants with Duchenne muscular dystrophy (DMD) (age 6 to <12 years).

DETAILED DESCRIPTION:
This is a global, randomized, double-blind, trial of pamrevlumab or placebo in combination with systemic corticosteroids in participants with DMD, aged 6 to <12 years (ambulatory participants only). Approximately 70 participants will be randomized at a 1:1 ratio to Arm A (pamrevlumab + systemic deflazacort or equivalent potency of corticosteroids administered orally) or Arm B (placebo+ systemic deflazacort or equivalent potency of corticosteroids administered orally), respectively. Randomization will be stratified by exon 44 deletion for analysis. Stratification has no impact upon treatment assignment nor dosage.

Participants must be fully informed of the potential benefits of approved products and make an informed decision when participating in a clinical trial in which they could be randomized to placebo.

The main study has 3 study periods:

* Screening period: Up to 4 weeks
* Treatment period: 52 weeks
* Safety Follow-up period/final assessment: A visit 28 days (+/- 3 Days) and a final safety follow-up phone call 60 days (+ 3 Days) after the last dose

Each participant will receive pamrevlumab or placebo at 35 mg/kg every 2 weeks for up to 52 weeks. Participants who complete 52 weeks of treatment may be eligible for an open-label extension (OLE), offering extended treatment with pamrevlumab.

Participants who discontinue study treatment for any reason should be encouraged to return to the investigative site to complete final safety and efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

Age, and consent:

1. Males at least 6 to <12 years of age at screening initiation
2. Written consent by participant and/or legal guardian as per regional/ country and/or Institutional Review Board (IRB)/Independent Ethics Committee (IEC) requirements

   DMD diagnosis:
3. Medical history includes diagnosis of DMD and confirmed Duchenne mutation, including status of exon 44 using a validated genetic test.

   Pulmonary criteria:
4. Average (of screening and Day 0) percent predicted forced vital capacity (FVC) above 45%
5. On a stable dose of systemic corticosteroids for a minimum of 6 months, with no substantial change in dosage for a minimum of 3 months (except for adjustments for changes in body weight) prior to screening. Corticosteroid dosage should be in compliance with the DMD Care Considerations Working Group recommendations (for example, prednisone or prednisolone 0.75 mg/kg per day or deflazacort 0.9 mg/kg per day) or stable dose. A reasonable expectation is that dosage and dosing regimen would not change significantly for the duration of the study.

   Performance criteria:
6. Able to complete 6-minute walking distance (6MWD) test with a distance of at least 270 meters but no more than 450 meters on two occasions within 3 months prior to randomization with ≤10% variation between these two tests.
7. Able to rise (TTSTAND) from floor in <10 seconds (without aids/orthoses) at screening visit.
8. Able to undergo magnetic resonance imaging (MRI) test for the lower extremities vastus lateralis muscle.

   Vaccination:
9. Agreement to receive annual influenza vaccinations during the conduct of the study.

   Laboratory criteria:
10. Adequate renal function: cystatin C ≤1.4 mg/liter (L)
11. Adequate hematology and electrolytes parameters:

    1. Platelets >100,000/microliter (μL)
    2. Hemoglobin >12 grams (g)/deciliter (dL)
    3. Absolute neutrophil count >1500/μL
    4. Serum calcium (Ca), potassium (K), sodium (Na), magnesium (Mg) and phosphorus (P) levels are within a clinically accepted range for DMD participants
12. Adequate hepatic function:

    1. No history or evidence of liver disease
    2. Gamma glutamyl transferase (GGT) ≤3x upper limit of normal (ULN)
    3. Total bilirubin ≤1.5xULN

Exclusion Criteria:

General Criteria:

1. Concurrent illness other than DMD that can cause muscle weakness and/or impairment of motor function
2. Severe intellectual impairment (for example, severe autism, severe cognitive impairment, severe behavioral disturbances) preventing the ability to perform study assessments in the Investigator's judgment
3. Previous exposure to pamrevlumab
4. Body mass index (BMI) ≥40 kg/square meter (m^2) or weight >117 kg
5. History of

   1. allergic or anaphylactic reaction to human, humanized, chimeric or murine monoclonal antibodies
   2. hypersensitivity to study drug or any component of study drug
6. Exposure to any investigational drug (for DMD or not), in the 30 days prior to screening initiation or use of approved DMD therapies (for example, eteplirsen, ataluren, golodirsen, casimersen) within 5 half-lives of screening, whichever is longer with the exception of the systemic corticosteroids, including deflazacort

   Pulmonary and Cardiac criteria:
7. Requires ≥16 hours continuous ventilation
8. Poorly controlled asthma or underlying lung disease such as bronchitis, bronchiectasis, emphysema, recurrent pneumonia that in the opinion of the investigator might impact respiratory function
9. Hospitalization due to respiratory failure within the 8 weeks prior to screening
10. Severe uncontrolled heart failure (New York Heart Association [NYHA] Classes III-IV) or renal dysfunction, including any of the following:

    1. Need for intravenous diuretics or inotropic support within 8 weeks prior to screening
    2. Hospitalization for a heart failure exacerbation or arrhythmia within 8 weeks prior to screening
    3. Participants with glomerular filtration rate (GFR) of less than 30 mL/minute (min)/1.73 m^2 or with other evidence of acute kidney injury as determined by investigator
11. Arrhythmia requiring anti-arrhythmic therapy
12. Any other evidence of clinically significant structural or functional heart abnormality

    Clinical judgment:
13. The Investigator judges that the participant will be unable to fully participate in the study and complete it for any reason, including inability to comply with study procedures and treatment, or any other relevant medical, surgical or psychiatric conditions

Ages: 6 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (27):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California Davis Children's Hospital, Sacramento, California
  - University of California San Diego Health, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Rare Disease Research - Tampa, Tampa, Florida
  - Rare Disease Research Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center Research Institute, Fairway, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Center, Worcester, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Spectrum Health Hospitals Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Shriners Hospital for Children, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia Children's Hospital, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Wisconsin Corporate Center, Milwaukee, Wisconsin
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Klinik Favoriten, Vienna, Vienna, Austria
- Belgium (3):
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Flemish Brabant
  - Centre Hospitalier Régional de la Citadelle, Liège, Liege
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
- London Health Sciences Centre, London, Ontario, Canada
- China (5):
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The 1st Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changsha, Hunan
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
- France (3):
  - Hôpital Hautepierre, Strasbourg, Bas-Rhin
  - Centre Hospitalier Universitaire Nantes - Hôtel Dieu, Nantes
  - Association Institut de Myologie, Paris
- Italy (5):
  - IRRCS Ospedale San Raffaele, Milan, Milan
  - Istituto di Ricovero e Cura a Carattere Scientifico Eugenio Medea - Lombardia, Bosisio Parini
  - Centro Clinico NeMO, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale Pediatrico Bambino Gesù - Roma - Gianicolo, Roma
- Netherlands (2):
  - Leiden Universitair Medisch Centrum, Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen
- Spain (2):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds, England
  - Oxford University Hospitals NHS Foundation Trust, Oxford, England

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included 2 periods: a Double-blind (DB) period and an Open-label extension (OLE) period.
Groups:
- Pamrevlumab: Participants received pamrevlumab 35 milligrams (mg)/kilogram (kg) by intravenous (IV) infusion every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks in the DB period and continued to receive the same dose of pamrevlumab for up to 52 weeks in the OLE period or until pamrevlumab was commercially available, or the sponsor decided to end the study, whichever occurred first.
- Placebo: Participants received placebo matched to pamrevlumab by IV infusion every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks in the DB period. Participants received pamrevlumab 35 mg/kg by IV infusion every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks in the OLE period or until pamrevlumab was commercially available, or the sponsor decided to end the study, whichever occurred first.
Period: DB Period (52 Weeks)
Arm/Group | Pamrevlumab | Placebo
Started | 37 | 36
Received at Least 1 Dose of Study Drug | 36 | 36
Completed | 35 | 36
Not Completed | 2 | 0
Not completed — Participant/Legal Guardian Decision | 2 | 0
Period: OLE Period (52 Weeks)
Arm/Group | Pamrevlumab | Placebo
Started | 34 (1 participant who completed DB period, did not roll over into the OLE period.) | 35 (1 participant who completed DB period, did not roll over into the OLE period.)
Received at Least 1 Dose of Study Drug | 34 | 34
Completed | 0 | 0
Not Completed | 34 | 35
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Participant/Legal Guardian Decision | 11 | 13
Not completed — Sponsor Decision to Terminate Study | 21 | 19
Not completed — Other than specified | 0 | 1
Not completed — Entered into OLE but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) set included all randomized participants.
Groups:
- Pamrevlumab: Participants received pamrevlumab 35 mg/kg by IV infusion every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks in the DB period and continued to receive the same dose of pamrevlumab for up to 52 weeks in the OLE period or until pamrevlumab was commercially available, or the sponsor decided to end the study, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Pamrevlumab | Placebo | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.46) | 9.0 (1.56) | 9.0 (1.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 37 | 36 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 34 | 28 | 62
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 9 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 23 | 22 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in North Star Ambulatory Assessment (NSAA) Total Score at Week 52
Description: The NSAA consisted of 17 activities, each scored as 0 (activity could not be performed), 1 (modified method but achieved goal without physical assistance from another), or 2 (normal, achieved goal without assistance). The sum of these 17 scores was used to form a total score ranging from 0 (worst) to 34 (fully independent function). If fewer than 15 of the 17 activities were performed, the total score was considered missing. If 15 to 16 activities were performed, the total score was calculated by multiplying the sum of the scores in the x activities that were performed by 17/x. If an activity could not be performed due to disease progression/loss of ambulation, a score of 0 was assigned. Higher scores indicated better functioning. Least square (LS) mean and standard error (SE) were analyzed using a mixed model for repeated measure (MMRM).
Time Frame: Baseline, Week 52
Population: The ITT set included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 36 | 36
units on a scale | -3.022 (0.5505) | -2.494 (0.6962)
Statistical Analysis 1: Comparison: Pamrevlumab vs Placebo; Test type: Other; p = 0.5553, Mixed Models Analysis; LS Mean Difference = -0.528, 95% CI 2-sided [-2.308 to 1.251], Standard Error of Mean 0.8912

2. Secondary Outcome: Change From Baseline in 4-Stair Climb Velocity (4SCV) Assessment at Week 52
Description: The 4SCV (centimeters [cm]/second [sec]) was calculated as the ratio of the total height (cm) of stairs climbed divided by the number of seconds taken to complete the 4-stair climb.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 36 | 36
cm/sec | -1.858 (4.5459) | -3.797 (5.1899)

3. Secondary Outcome: Change From Baseline in the 10-Meter Walk/Run Test at Week 52
Description: The time (in sec) required for a participant to run or walk a distance of 10 meters as quickly as possible was calculated as velocity (meters/sec).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/sec
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 36 | 36
meters/sec | -0.176 (0.2193) | -0.196 (0.3552)

4. Secondary Outcome: Change From Baseline in Time to Stand (TTSTAND) at Week 52
Description: The time (in sec) required for a participant to stand from supine position has been reported. A longer time taken reflected a worse outcome.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 36 | 31
sec | 2.24 (3.353) | 1.94 (3.688)

5. Secondary Outcome: Time to Loss of Ambulation (LoA) From Baseline to Week 52
Description: Time (days) to LoA was defined as the number of days from randomization to the date of LoA, or all-cause death based on observed data, whichever occurred earlier during the on-study period. Median time (days) to LoA was calculated using Kaplan Meier Survival Estimates.
Time Frame: Baseline to Week 52
Population: The ITT set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 37 | 36
days | NA [NA to NA] — Due to insufficient number of participants with an event of LoA or death, median and 95% confidence interval (CI) could not be calculated. | NA [NA to NA] — Due to insufficient number of participants with an event of LoA or death, median and 95% CI could not be calculated.

ADVERSE EVENTS:
Time Frame: Baseline up to Week 129
Description: As pre-specified, All-cause mortality data were collected and reported for all enrolled participants; and Serious and Non-serious adverse events data were collected and reported for all participants who received any dose of study medication.
Groups:
- DB Period: Pamrevlumab: Participants received pamrevlumab 35 mg/kg by IV infusion every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks in the DB period.
- DB Period: Placebo: Participants received placebo matched to pamrevlumab by IV infusion every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks in the DB period.
- OLE Period: Pamrevlumab: Participants received pamrevlumab 35 mg/kg by IV infusion every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks in the OLE period or until pamrevlumab was commercially available, or the sponsor decided to end the study, whichever occurred first.
Arm/Group | DB Period: Pamrevlumab | DB Period: Placebo | OLE Period: Pamrevlumab
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/36 | 0/69
Serious Adverse Events (participants affected / at risk) | 3/36 | 1/36 | 0/68
Other Adverse Events (participants affected / at risk) | 35/36 | 33/36 | 45/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Pamrevlumab (N=36) | DB Period: Placebo (N=36) | OLE Period: Pamrevlumab (N=68)
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Pamrevlumab (N=36) | DB Period: Placebo (N=36) | OLE Period: Pamrevlumab (N=68)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 3 | 6
Nausea (Gastrointestinal disorders) | 2 | 3 | 4
Vomiting (Gastrointestinal disorders) | 10 | 7 | 12
Fatigue (General disorders) | 4 | 5 | 2
Gait disturbance (General disorders) | 0 | 2 | 0
Injection site bruising (General disorders) | 0 | 2 | 1
Pyrexia (General disorders) | 9 | 7 | 10
COVID-19 (Infections and infestations) | 16 | 8 | 4
Ear infection (Infections and infestations) | 1 | 4 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 3
Influenza (Infections and infestations) | 2 | 1 | 4
Nasopharyngitis (Infections and infestations) | 10 | 7 | 11
Pharyngitis (Infections and infestations) | 2 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 8 | 6
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 2 | 3
Joint injury (Injury, poisoning and procedural complications) | 3 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 3 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Vascular access site pain (Injury, poisoning and procedural complications) | 1 | 2 | 0
Blood pressure diastolic decreased (Investigations) | 2 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3
Headache (Nervous system disorders) | 14 | 5 | 5
Hypokinesia (Nervous system disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT04632940/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT04632940/SAP_001.pdf